CLINICAL TRIAL: NCT05217277
Title: Clinical and Biochemical Evaluation of Dental and Periodontal Conditions in Children With Juvenile Idiopathic Arthritis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-146
Record Dates: First submitted 2022-01-21; First posted 2022-02-01 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-01

CONDITIONS: Juvenile Idiopathic Arthritis; Gingivitis; Decay, Dental
Keywords: pediatric dentistry; periodontal status; juvenile idiopathic arthritis
MeSH Terms: conditions — Arthritis, Juvenile; Gingivitis; Dental Caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- patient with juvenile idiopathic arthritis and gingivitis: It is a group of patients between the ages of 5 and 16 who have recently been diagnosed with juvenile idiopathic arthritis and gingivitis, have not used medication yet.
  Interventions: Diagnostic Test: Humans ELISA kits
- healthy patient group with gingivitis: It is a group of healthy patients with gingivitis between the ages of 5-16 who have not taken antibiotics in the last 3 months.
  Interventions: Diagnostic Test: Humans ELISA kits
- healthy patient group without gingivitis: It is a group of healthy patients without gingivitis between the ages of 5-16 who have not taken antibiotics in the last 3 months.
  Interventions: Diagnostic Test: Humans ELISA kits
- patient with juvenile idiopathic arthritis and without gingivitis: It is a group of patients between the ages of 5 and 16 who have recently been diagnosed with juvenile idiopathic arthritis and without gingivitis, have not used medication yet.
  Interventions: Diagnostic Test: Humans ELISA kits

INTERVENTIONS:
Diagnostic Test: Humans ELISA kits — ELISA (enzyme-linked immunosorbent assay) is a plate-based assay technique designed for detecting and quantifying soluble substances such as peptides, proteins, antibodies, and hormones.
  The saliva of the patients included in the study will be examined with ELISA kits after they are taken.

SUMMARY:
Aimed to be done in the planned thesis to evaluate the dental and periodontal health of patients with newly diagnosed JIA and healthy-periodontal problems with cytokines from saliva and oxidative stress markers non-invasively, and thus, to determine the markers' evaluability in terms of markers in determining the state of inflammation among individuals with and without the disease.

DETAILED DESCRIPTION:
Periodontal diseases and inflammatory diseases such as arthritis show similar clinical pathologies such as connective tissue deterioration and bone destruction. They carry the risk of being seen together and the possibility of mutual influence. It is important whether these patients have a difference in cytokine profile from individuals who do not have the disease. In the literature, it has been determined that pro and anti-inflammatory cytokines, which are involved in the pathogenesis of periodontitis, are also involved in the pathogenesis of juvenile idiopathic arthritis (JIA). Cytokines play an undeniable role in the pathogenesis of both diseases. The cytokine profile in periodontal disease is distinctly similar to that of rheumatoid arthritis (RA). As in RA, the level of pro-inflammatory cytokines such as interleukin-1 beta (IL-1β) and tumor necrosis factor-alpha (TNF-α) increase in periodontal disease. Again, it is stated that oxidative stress assessment is an important factor in evaluating the development of the disease. Saliva evaluation can be made with new oxidative stress markers that can be used in this sense.

On the subject of the proposed thesis; It is to determine the profile of dental and periodontal health in a specific group in terms of biochemical and microbiology using different body fluids together with clinical findings and has an interdisciplinary character. Aimed to be done in the planned thesis;

It was aimed to evaluate the dental and periodontal health of patients with newly diagnosed JIA and healthy-periodontal problems with cytokines from saliva and oxidative stress markers non-invasively, and thus, to determine the markers' evaluability in terms of markers in determining the state of inflammation among individuals with and without the disease.

ELIGIBILITY:
Inclusion Criteria:

* healty patients

Exclusion Criteria:

* used antibiotics within the last 3 months

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients who have no disease other than juvenile idiopathic arthritis, newly diagnosed and not yet using medication.
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2020-05-06 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
biochemical evaluation of saliva in juvenile idiopathic arthritis | baseline
  Saliva samples were taken from the patients and the levels of interleukin-17, TNF alpha and Total antioxidant status in the saliva were measured with ELISA kits.

SECONDARY OUTCOMES:
Evaluation of oral hygiene in patients with juvenile idiopathic arthritis | baseline
  The number of caries in the patient was evaluated with the DMFT-dft index.
Evaluation of periodontal health in patients with juvenile idiopathic arthritis | baseline
  Silness-Loe plaque index (PI) was used to assess periodontal health.
Examination of periodontal health in patients with juvenile idiopathic arthritis | baseline
  Gingival index (GI) was also used to examination periodontal health.
periodontal health in patients with juvenile idiopathic arthritis | baseline
  Bleeding on prob index were used for periodontal health examination.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Sozeri, Study Chair — researcher; Ferhat Demir, Study Chair — researcher; Selin Yıldırım, Study Chair — researcher
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Maltepe, Turkey (Türkiye)